CLINICAL TRIAL: NCT06038318
Title: Promoting Resilience in Early Survivorship Among Adolescents and Young Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Abby Rosenberg, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-652; R01CA269574-01 (NIH)
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Stress; Anxiety
Keywords: Stress Management
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRISM Program Mobile App (Experimental): Participants will be randomized to "app-only" group and will complete:
  * Baseline questionnaire.
  * mPRISM App self guided modules
  * 3 month questionnaire.
  * mPRISM App self guided modules until final survey at 6 months and end of participation.
  Interventions: Behavioral: mPRISM Program App
- PRISM Program Video Coach (Active Comparator): Participants will be randomized to "video" group and will complete:
  * Baseline questionnaire.
  * PRISM sessions.
  * 3 month questionnaire with re-randomization to either "app-only" or "text" groups or referral to specialty psychosocial support.
  * After re-randomization, participants will complete PRISM sessions until final survey at 6 months and end of participation.
  Interventions: Behavioral: PRISM Program Video Coach; Behavioral: mPRISM Program App
- PRISM Program Text Coach (Active Comparator): Participants will be randomized to "text" group and will complete:
  * Baseline questionnaire.
  * PRISM sessions.
  * 3 month questionnaire with re-randomization to "app-only," "text," or "video" groups.
  * After re-randomization, participants will complete PRISM sessions until final survey at 6 months and end of participation.
  Interventions: Behavioral: PRISM Program Text Coach; Behavioral: mPRISM Program App

INTERVENTIONS:
Behavioral: PRISM Program Video Coach — A 6-session, skills-based, manualized resilience education program delivered via video coaching by trained English or Spanish speaking PRISM coaches. Participants will have complete access to the PRISM Program mobile app. Sessions will be delivered by a HIPAA compliant videoconferencing platform, Zoom, approximately every 1-2 weeks based on participant preference. For participants who do not have smartphones, temporary equipment will be provided.
  Other Names: Promoting Resilience in Stress Management
  Arms: PRISM Program Video Coach
Behavioral: PRISM Program Text Coach — A 6-session, skills-based, manualized, resilience education program delivered via text coaching by trained English or Spanish speaking PRISM coaches. Participants will have complete access to the PRISM Program mobile app. Sessions will be delivered by HIPAA compliant SMS text-messaging service, Zoom, approximately every other week. For participants who do not have smartphones, temporary equipment will be provided.
  Other Names: Promoting Resilience in Stress Management
  Arms: PRISM Program Text Coach
Behavioral: mPRISM Program App — 6 static modules to practice skills-based, manualized, resilience education program delivered via PRISM Program mobile app. For participants who do not have smartphones, temporary equipment will be provided.
  Other Names: Promoting Resilience in Stress Management

SUMMARY:
The goal of this study is to find the best way to help participants and families manage the stress of facing a serious illness and be better able to "bounce back" or be resilient after a difficult situation. Participants will take part in the "Promoting Resilience in Stress Management" PRISM program, which is designed to provide skills to change or improve the impact of stress in everyday life.

The name of the intervention used in this research study is:

-PRISM (a mobile app program comprised of 6 sessions of skills-based, manualized resilience education)

DETAILED DESCRIPTION:
In this sequential, multiple assignment, randomized trial participants will be randomly selected to participate in PRISM program sessions with a trained research coach either by text or by video sessions, or participants will use the PRISM mobile app program in a self-guided way. Randomization means the group participants are placed in will be decided by chance. All groups will continue to receive all the same care from primary medical, social work, and other care teams.

In this two-stage study, participants will be randomly assigned to either the "app-only" (20% chance), "text" (40% chance) or "video" (40% chance) groups for the first stage. In the second stage, participants may be re-randomized again to the "app-only," or "text," groups, or will be referred to a specialty psychosocial support, social worker or counselor, based on responses to questionnaires. Participants randomized to the "app-only" group in the first stage will not be re-randomized.

The research study procedures include screening for eligibility and completion of questionnaires.

Participation in this research study is expected to last for up to 6 months.

It is expected about 325 people will take part in this research study.

The National Institute for Health (NIH) is funding this research study.

ELIGIBILITY:
Participants that have completed their main cancer-directed therapy at one of the study sites affiliated centers who meet all the eligibility criteria will be eligible for participation in this study.

Inclusion Criteria:

* All genders ≥ 12 and ≤ 25 years of age at baseline
* Participant is able to speak English or Spanish language (for PRISM sessions)
* Participant is able to read English or Spanish language (for completion of surveys)
* Participant is cognitively able to participate in PRISM sessions and complete written questionnaires and surveys, as judged by the site investigator

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 325 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Connor Davidson Resilience Scale (CDRISC-10) Score | At 6 months
  Assessed by the CDRISC-10, a 10-item measures consisting of a 5-point Likert scale with answers ranging from 0 (not true at all) to 4 (true nearly all the time) for a total of 40 points. Higher scores reflect greater resilience. Evaluation will be based on the scores of the video and text cohorts vs. the self-guided cohort.

SECONDARY OUTCOMES:
CDRISC-10 Score for App-Only Cohort Responders | 3 months
  Assessed by the CDRISC-10, a 10-item measures consisting of a 5-point Likert scale with answers ranging from 0 (not true at all) to 4 (true nearly all the time) for a total of 40 points. Higher scores reflect greater resilience. Participant "responders" are defined as having sustained CDRISC scores >29 after PRISM sessions or increased by >2 points at the timepoints.
CDRISC-10 Score for Text Coach Cohort Responders | 3 months
  Assessed by the CDRISC-10, a 10-item measures consisting of a 5-point Likert scale with answers ranging from 0 (not true at all) to 4 (true nearly all the time) for a total of 40 points. Higher scores reflect greater resilience. Participant "responders" are defined as having sustained CDRISC scores >29 after PRISM sessions or increased by >2 points at the timepoints.
Change in HOPE Scale Score | At Baseline, 3 months, and 6 months
  Assessed by the HOPE Scale, a 12-item measures scored on an 8-point Likert scale with answers ranging from 1 "Definitely False" to 8 "Definitely True" for a total score of 96. A higher score implies a greater level of hopeful thought patterns.
Change in Adolescent Participant Quality of Life Total Score | At Baseline, 3 months, and 6 months
  Assessed by the Pediatric Quality of Life (PedsQL) Generic Core Scales Short Form (SF15) (Teen or Child Report) and PedsQL Cancer Module (Child or Teen Report) scales, 42-items to evaluate health-related quality of life. Items are rated on a 5-point Likert scale with answers ranging from 0 "Never" to 4 "Almost Always" for a score range of 0 - 100. A higher score represents better health-related quality of life.
Change in Young Adult Participant Quality of Life Total Score | At Baseline, 3 months, and 6 months
  Assessed by the Pediatric Quality of Life (PedsQL) Generic Core Scales Short Form (SF15) Young Adult Report and PedsQL Cancer Module Young Adult Report scales, 42-items to evaluate health-related quality of life. Items are rated on a 5-point Likert scale with answers ranging from 0 "Never" to 4 "Almost Always" for a score range of 0 - 100. A higher score represents better health-related quality of life.
Change in Kessler-6 Psychological Distress Scale Score | At Baseline, 3 months, and 6 months
  Assessed by the Kessler-6, a 6-item measure for the level of psychological distress in the past month. Responses are scored on a 5-point Likert scare with answers ranging from 0 "None of the time" to 4 "All of the time," and with a total score range of 0 - 4. Scores > or = 7 suggest "high" distressed and those > or = 13 meet criteria for serious or debilitating psychological distress.
Change in Hospital Anxiety and Depression Scale (HADS) Anxiety Subscale Score | At Baseline, 3 months, and 6 months
  Assessed by the HADS-A subscale which is comprised of 7 items. Items are scored 0-3 with a subscale total score range of 0 - 21. A higher scores represents increasing abnormality (or caseness) for anxiety.
Change in HADS Depression Subscale Score | At Baseline, 3 months, and 6 months
  Assessed by the HADS-D subscale score which is comprised of 7 items. Items are scored 0-3 with a subscale total score range of 0 - 21. A higher score represents increasing abnormality (or caseness) for depression.

CONTACTS AND LOCATIONS:
Overall Officials: Abby Rosenberg, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu